CLINICAL TRIAL: NCT00688805
Title: Effects of Propranolol on Responses to Drug-Related Imagery Scripts
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Basic Science
Other Study IDs: 999908433; 08-DA-N433
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-12-16

CONDITIONS: Cocaine Dependence
Keywords: Propanolol; Substance Abuse; Craving; Imagery; Drug Cues; Cocaine
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Propranolol

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Propranolol
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — 40 mg given as a single oral administration in an opaque capsule
  Arms: Arm 1
Drug: Placebo — matching capsule containing no active medication
  Arms: Arm 2

SUMMARY:
Background:

* Relapse to drug abuse is thought to result, in many cases, from exposure to cues that trigger drug-related memories or emotional associations for example, the association between the sight of a crack pipe and a set of responses such as rapid heartbeat and desire for cocaine. This type of memory is reconsolidated (actively re-stored) each time it is reactivated; however, the reconsolidation process can be disrupted by the drug propranolol, which weakens the link between that memory and an emotional response.
* Propranolol is traditionally used to treat high blood pressure and other heart-related conditions. Researchers are interested in studying whether propranolol disrupts reconsolidation of drug-cued memories in individuals who are addicted to cocaine.

Objectives:

- To examine whether propranolol can interfere with reconsolidation of cocaine-related memories and reduce cravings and drug use in substance abusers.

Eligibility:

- Individuals between 18 and 55 years of age who are current cocaine users enrolled in a methadone treatment program.

Design:

* The study will involve four long sessions (visits 1, 4, 6, and 14) and 10 short sessions. The short visits will be for monitoring of participants use of drugs and alcohol; the longer visits will involve more tests and lab sessions. Participants will be randomized to either the propranolol or placebo group.
* The long sessions will involve the following procedures:
* An interview session to develop a personalized drug script/cue set.
* A two-hour intervention session with baseline measures, drug administration (propranolol or placebo), and two script-guided imagery sets. This is the only administration of propranolol during the study.
* Two follow-up test sessions, 1 and 5 weeks after the intervention session.
* Participants will make brief visits to our outpatient clinic for twice-weekly monitoring of ongoing drug use via urine screens and self-report, starting 1 week before the intervention session and ending 5 weeks later.

DETAILED DESCRIPTION:
Background

Relapse to drug abuse or addiction is thought to result, in many cases, from exposure to cues that elicit drug-related memories. The term memories is used here not in its everyday sense, but in a sense that corresponds more closely to emotional associations for example, the association between the sight of a crack pipe and a set of responses such as rapid heartbeat and desire for cocaine. Studies in rodents and humans show that this type of memory is reconsolidated (actively re-stored) each time it is reactivated, and that the reconsolidation process can be disrupted by propranolol. Such disruption does not erase the autobiographical memory of an event, but instead weakens the link between that memory and an emotional response. Human studies are needed to determine whether propranolol disrupts reconsolidation of drug-cued memories in addicted individuals; this would present a novel and exciting therapeutic possibility for preventing craving and relapse.

Objective

To examine whether administration of propranolol interferes with reconsolidation of cocaine-related memories and reduces cravings and drug use in substance abusers.

Study population

Up to 200 (60 evaluable) individuals maintained on methadone and using cocaine will be recruited from local treatment programs. The target enrollment will include 40% women and 60% minorities.

Experimental design and methods

Participants will be randomized to one of two groups: propranolol (40 mg, oral, immediate-release formulation) or placebo. The study will include four laboratory sessions: (1) An information-gathering session that includes an interview to obtain information for development of a personalized drug script/cue set. (2) A two-hour intervention session in which there will be baseline measures, drug administration (propranolol or placebo, double blind), and, starting 60 min after drug administration, two script-guided imagery sets. Cue-responsivity data will be collected, but the main purpose of the session is interventional. This will be the only administration of propranolol during the study. (3, 4) Two follow-up test sessions, 1 and 5 weeks after the intervention session; participants responses to re-exposure to the personalized drug script/cue set will be measured. In addition to attending the four laboratory sessions, participants will make brief visits to our outpatient clinic for twice-weekly monitoring of ongoing drug use via urine screens and self-report, starting 1 week before the intervention session and ending 5 weeks later.

Outcome measures

Outcome measures will include subjective ratings of drug craving, autonomic responses (heart rate, blood pressure, galvanic skin response), and cocaine and heroin use (urine drug screens and self-reported drug use).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. - Age between 18 and 55 years
  2. - Evidence of current cocaine use (self-report)
  3. - Minimum lifetime cocaine use of one year (self-report)
  4. - Minimum use of cocaine of once in the past 30 days (self-report)
  5. - Enrolled in methadone maintenance

EXCLUSION CRITERIA:

1. - Allergy or hypersensitivity to propranolol or other beta blockers.
2. - History of: schizophrenia (or of any other DSM-IV psychotic disorder), anxiety disorders (e.g., panic disorder), or bipolar disorder.
3. - Current major depressive disorder.
4. - Current physical dependence on, or current abuse of, alcohol, benzodiazepines, or other sedative-hypnotic drugs.
5. - Cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires.
6. - Pregnant; breast feeding.
7. - Impaired hepatic function with AST or ALT greater than 5x the upper limit of normal.
8. - Medical conditions that would contraindicate administration of propranolol (e.g., uncompensated congestive heart failure; pulmonary edema; asthma; COPD; history of severe allergic reactions (seasonal, environmental, food, medications, etc.); Raynaud s disease; second- or third-degree atrioventricular block; arrhythmias other than sinus arrhythmia; thyroid dysfunction; diabetes mellitus; renal impairment.

   Per the American Thoracic Society (ATS), COPD Clinical assessment is based on medical history and physical examination. Although a complete examination is indicated for all patients, these two components are specifically important for patients with suspected COPD. (ATS & ERS, 2004) Accordingly, if medical history and physical exam suggest possible COPD the participant will be forwarded for spirometry/pulmonary function tests to aid in the diagnosis.
9. - Bradycardia (heart rate < 60 bpm) on three consecutive readings.
10. - Systolic blood pressure < 100 mm Hg; diastolic blood pressure < 60 mm Hg; on three consecutive readings.
11. - Medications that could interact with propranolol either pharmacodynamically or pharmacokinetically to produce adverse effects. Such medication would include CNS depressants (e.g., barbiturates, benzodiazepines, other sedatives), antihypertensive medications (including nitrates), antiarrhythmic medications, antiseizure medications (dilantin), acetylcholinesterase inhibitors (e.g., donepezil, galantamine), aminoquinolines (antimalarial), antipsychotic medications, beta agonists, insulin, MAOIs, NSAIDs, rifamycin derivatives, rizatriptan, SSRIs, sulfonylureas, theophylline, pseudophedrine, phenylephrine, ephedrine, epinephrine, noriepinephrine, amphetamines, and some herbal supplements.
12. - Current use of beta blockers for any medical condition.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-12-12; Primary Completion 2013-12-16 (Actual); Study Completion 2013-12-16 (Actual)

PRIMARY OUTCOMES:
Drug craving | 1 hr

SECONDARY OUTCOMES:
Galvanic skin response | 1 hr

CONTACTS AND LOCATIONS:
Overall Officials: Kenzie Preston, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Abduljawad KA, Langley RW, Bradshaw CM, Szabadi E. Effects of clonidine and diazepam on the acoustic startle response and on its inhibition by 'prepulses' in man. J Psychopharmacol. 1997;11(1):29-34. doi: 10.1177/026988119701100110. PMID 9097890
- [Background] Benschop RJ, Jacobs R, Sommer B, Schurmeyer TH, Raab JR, Schmidt RE, Schedlowski M. Modulation of the immunologic response to acute stress in humans by beta-blockade or benzodiazepines. FASEB J. 1996 Mar;10(4):517-24. doi: 10.1096/fasebj.10.4.8647351.
- [Background] Berger SP, Hall S, Mickalian JD, Reid MS, Crawford CA, Delucchi K, Carr K, Hall S. Haloperidol antagonism of cue-elicited cocaine craving. Lancet. 1996 Feb 24;347(9000):504-8. doi: 10.1016/s0140-6736(96)91139-3. PMID 8596268